CLINICAL TRIAL: NCT01371682
Title: An Open Label Study Conducted in Healthy Subjects to Demonstrate Bioequivalence Between Ropinirole Prolonged Release Tablets (Ropinirole XL, Marketed as REQUIP-MODUTAB™, REQUIP XL™ at 2 mg) Manufactured at Crawley and Aranda
Brief Title: A Study Conducted in Healthy Subjects to Demonstrate Bioequivalence Between Ropinirole Prolonged Release Tablets Manufactured at Crawley and Aranda
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 112771
Record Dates: First submitted 2010-06-10; First posted 2011-06-13 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Session 1 (Other): Ropinirole manufactued at Crawley will be compared to that manufactured at Aranda
  Interventions: Drug: Ropinirole XL
- Session 2 (Other): Ropinirole manufactured at Crawley will be compared to that manufactured at Aranda.
  Interventions: Drug: Ropinirole XL

INTERVENTIONS:
Drug: Ropinirole XL — Ropinirole XL manufactured at Crawley will be compared to that manufactued at Aranda.

SUMMARY:
This is an open-label, randomised, two-period crossover, single dose study to demonstrate bioequivalence between the extended release 2 mg ropinirole XL tablets manufactured at two different sites in healthy subjects. Dosing will be under fasting conditions and there will be a minimum one week washout between doses. Domperidone will be administered to control dopaminergic side effects. Pharmacokinetic samples will be taken following each dose. Safety assessments will include screening and follow-up vital signs, ECGs and safety laboratory tests. Vital signs and adverse events will be monitored periodically throughout the study.

DETAILED DESCRIPTION:
This is an open-label, randomised, two-period crossover, single dose study to demonstrate bioequivalence between the extended release 2 mg ropinirole XL tablets manufactured at two different sites in healthy subjects. Dosing will be under fasting conditions and there will be a minimum one week washout between doses. Domperidone will be administered to control dopaminergic side effects. Pharmacokinetic samples will be taken following each dose. Safety assessments will include screening and follow-up vital signs, ECGs and safety laboratory tests. Vital signs and adverse events will be monitored periodically throughout the study.

The manufacturing of ropinirole XL tablets will be moved from the Crawley (UK) manufacturing facility to the Aranda (Spain) manufacturing facility. The tablets manufactured at Aranda will have the same characteristics as those manufactured at Crawley.

The present pharmacokinetic study is designed to assess bioequivalence of ropinirole XL 2 mg tablets manufactured at Aranda vs ropinirole XL 2 mg tablets manufactured at Crawley. Bioequivalence between the two tablets will be tested in healthy subjects and administered in the fasting state.

ELIGIBILITY:
* Inclusion Criteria
* Male or female healthy subjects aged between 18 and 50 years of age inclusive at dosing.
* Body mass index of 19 to 30 kg/m2, with a body weight of at least 50 kg.
* No abnormality on clinical examination.
* No abnormality revealed by the clinical chemistry or haematology examination at the pre study medical examinationA normal 12 lead ECG at the pre study screening.
* QTc interval of < 450msec at screening.
* Normal systolic (100 140mmHg) and diastolic (<90mmHg) blood pressure (supine) at pre study screening.
* AST, ALT and alkaline phosphatase within the laboratory reference range and bilirubin £ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Subjects must have provided written informed consent prior to performing any assessments.A female subject is eligible to participate if she is of:Choose one or both of criteria below depending on requirements of study:Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Since co-administration of HRT with ropinirole has been shown to decrease the clearance of ropinirole, subjects on hormone replacement therapy (HRT) will be excluded.Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to continue using the same method of contraception until at least one month after completion of the study (i.e. one month after the follow-up visit).
* Male subjects must agree to use one of the contraception methods
* Exclusion criteria
* Any clinically relevant abnormality identified on the screening history and physical or laboratory examination or any other medical condition or circumstance making the volunteer unsuitable for participation in the study
* Definite or suspected personal history or family history of adverse reactions or hypersensitivity to the study drug or to drugs with a similar chemical structure or to domperidone or a personal history of lactose intolerance.
* History or presence of clinically significant cardiovascular, neurological, psychiatric, haematological or renal abnormalities.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of surgical procedures that might affect the absorption of ropinirole (e.g., partial/total gastrectomy, cholecystectomy).
* The subject has received prescription drugs within 14 days or 5 half-lives (whichever is longer) or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study or compromise safety.
* Systolic BP > 140 mm Hg and/or Diastolic BP > 90 mm Hg at screening or pre-dose.
* A history of moderate or severe dizziness, syncope, or orthostatic hypotension, defined as a fall in blood pressure after rising from the supine to erect posture, of >/= 30 mmHg for systolic pressure and >/= 20 mmHg for diastolic pressure at screening.
* History of excessive regular alcohol consumption within 6 months of screening defined as An average weekly intake of >21 units for males or > 14 units for females. One unit is equivalent to a half-pint (220mL) of beer, 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* Subjects who smoke >20 cigarettes per day and those who will not abstain from smoking or maintain a constant smoking habit for 14 days before dosing until 72 hours after the last dose.
* Positive urine drug screen (UDS) including alcohol and cotinine (for non-smokers) at screening or pre-dose visits.
* Positive hepatitis B virus, hepatitis C virus or Human Immunodeficiency Virus (HIV) test at screening. If documented negative test results have been obtained within the last 2 months, it will not be necessary to repeat these tests.
* Positive serum or urine beta-human chorionic gonadotropin (b-hCG) test (females).
* Women who are pregnant, lactating, or planning to become pregnant.
* Female subjects not willing to use proposed contraceptive methods (see Section 8.1.1).
* Female subjects taking hormone replacement therapy.
* Male subjects who are not willing to abstain from sexual intercourse or use a condom during sexual intercourse with pregnant or lactating females. Male subjects not willing to use adequate method of contraception (see Section 8.1.2) if engaging in sexual intercourse with a female who could become pregnant.
* Donation of blood in excess of 500 mL within 56 days prior to first dose of study medication.
* History of sensitivity to heparin, heparin-induced thrombocytopenia.
* Abnormal 12-lead ECG findings include, but are not limited to, the following: myocardial ischemia, clinically significant conduction abnormalities, or clinically significant arrhythmias. QTc (machine read) > 450 msec on the screening ECG.
* Subjects have had treatment with a new molecular entity (investigational drug) or any other trial during the previous 30 days or five half-lives, whichever is longer. (the washout is from last dose of study medication in the previous study until the first dose of study medication).
* Current evidence of drug abuse or history of drug abuse within one year of enrollment.
* Inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
* Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study.
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.
* Vulnerable subjects (e.g. persons kept in detention).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09-18 (Actual); Primary Completion 2009-12-02 (Actual); Study Completion 2009-12-02 (Actual)

PRIMARY OUTCOMES:
PK samples will be measured for each formulation and compared between sites. The units of measure for this will include PK parameters, for example, Bioavailability, clearance and volume of distribution and Area under the curve. | 6 months
  PK parameters used to measure this change : AUC(0-infinity), AUC(0-t), Cmax, tmax, lambda - z and t1/2

SECONDARY OUTCOMES:
Safety values including Vital signs, BP, ECG values will be taken from the study for each cohort dosed with each formulation. The change in values will be compared from each formulation and any change bewteeen the two cohorts will be examined. | 6 months
  BP measures will a Systolic BP &; Diastolic BP (Hg mm). ECG levels will be taken looking at QTc measures. Vital signs will include blood pressur and pulse rate will be recorded at pre-dose and at 1, 2, 4, 6, 12 and 24 hours post-dose of ropinirole

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] GSK has concluded that it is not feasible to publish this study in a peer-reviewed scientific journal because the nature of the study is unlikely to be of interest to a journal. GSK is providing the attached study results summary.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 112771 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112771?search=study&search_terms=112771#rs
- Available data/document: Dataset Specification: 112771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register